CLINICAL TRIAL: NCT07262541
Title: Assessment of Airway Opening Pressure in Invasively Ventilated Children
Acronym: AOP-KID
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP250763; ID-RCB Number : 2025-A01008-41 (Other: Agence nationale de sécurité du médicament et des produits de santé, France)
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-09

CONDITIONS: Acute Respiratory Distress Syndrome in Children
Keywords: Acute respiratory distress syndrome; Invasively ventilated children; Airway opening pressure (AOP) detection; Children
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Measurement of airway opening pressure with pediatric slow flow method on first (Experimental): Measurement of airway opening pressure in invasively ventilated pediatric patients with "pediatric slow flow method" on first and "fixed flow method" in a second time.
  Interventions: Other: Measurement of airway opening pressure
- Measurement of airway opening pressure with fixed flow method on first (Experimental): Measurement of airway opening pressure in invasively ventilated pediatric patients with "fixed flow method" on first and "pediatric slow flow method" in a second time.
  Interventions: Other: Measurement of airway opening pressure

INTERVENTIONS:
Other: Measurement of airway opening pressure — Measurement of airway opening pressure in invasively ventilated pediatric patients with 2 methods, "fixed flow method" and "pediatric slow flow method". The two methods will be separated by a washout period. The order of the airway opening pressure detection methods will be random.

SUMMARY:
Acute respiratory distress syndrome (ARDS) in children is associated with significant morbidity and mortality. Current studies seek to individualize the management of children by defining several phenotypes, based until now mainly on clinical presentation. A better understanding of the respiratory mechanics of each patient could allow the individualization of other phenotypes and adapt their management with individualized ventilation. The method for detecting airway opening pressure (AOP) in children has not yet been validated and the reference methods in adults are difficult to apply in children due to their physiological particularities.

The main objective of the study is to evaluate the feasibility of two methods for measuring airway opening pressure in invasively ventilated pediatric patients.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) in children is associated with significant morbidity and mortality. Current studies seek to individualize the management of children by defining several phenotypes, based until now mainly on clinical presentation. A better understanding of the respiratory mechanics of each patient could allow the individualization of other phenotypes and adapt their management with individualized ventilation. The method for detecting airway opening pressure (AOP) in children has not yet been validated and the reference methods in adults are difficult to apply in children due to their physiological particularities.

The main objective of the study is to evaluate the feasibility of two methods for measuring airway opening pressure in invasively ventilated pediatric patients: "pediatric slow flow method" based on a recent bench study and "fixed flow method" based on an adult study. The two methods will be separated by a wash out.

The method will be considered feasible if at least one on three measures can be interpretated.

Air flow will be recorded using a pneumotachograph connected to a T piece.

ELIGIBILITY:
Inclusion Criteria:

* Minor patients aged > 1 year hospitalized in the pediatric intensive care unit at Necker-Enfants Malades Hospital and receiving invasive ventilation. To assess patients with acute respiratory distress syndrome, the PALICC-2 criteria are used.
* Holders of parental authority must be informed and consent to their child's participation in the study.
* The patient must be passively ventilated to ensure reliable measurements. This means that the patient must not be spontaneously ventilating and must be completely passively ventilated by the ventilator (no respiratory effort during long-term inflation).

Exclusion Criteria:

* Respiratory mechanics preventing interpretation of maneuvers (flow too low and/or resistance too high)
* Patient < 10 kg and/or child under 1 year of age
* Refusal by those with parental authority
* Patient not affiliated with social security
* Patient receiving AME (Medical Aid for Life)
* Contraindication or impossibility of performing static respiratory mechanics measurements: pneumothorax or pleural leak, head trauma or threatening HTIC, unstable patient with SpO2 < 88%, patient receiving nitric oxide (NO) (circuit leaks) or other circuit leaks or patient leaks > 20% displayed on the ventilator

Ages: 1 Year to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2031-01 (Estimated); Study Completion 2031-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of the two methods of measuring airway opening pressure | 5 years
  The method will be considered feasible if at least one maneuver out of three allows a measurement of the airway opening pressure to be obtained.

SECONDARY OUTCOMES:
Prevalence of airway opening pressure | 5 years
  Estimation of the prevalence of airway opening pressure during pediatric acute respiratory distress syndrome.
Value of airway opening pressure with each of the two measurement methods | 1 day
  Value of airway opening pressure with each of the two measurement methods of the study
Value of Positive end-expiratory pressure settled by the clinican and measured airway opening pressure | 1 day
  Value of Positive end-expiratory pressure settled by the clinican and measured airway opening pressure
Description of the tolerance of the two methods of measuring airway opening pressure | 5 years
  Description of the tolerance of the two methods of measuring airway opening pressure using the following parameters: minimum SpO2 value (%), variations in heart rate (HR, /min), systolic ans diastolic blood pressure (mmHg), expired CO2 (mmHg).
Duration of the methods | 5 years
  Duration of each method

CONTACTS AND LOCATIONS:
Overall Officials: Charlotte Collignon, M.D., Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Necker-Enfants Malades, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haudebourg AF, Moncomble E, Lesimple A, Delamaire F, Louis B, Mekontso Dessap A, Mercat A, Richard JC, Beloncle F, Carteaux G. A novel method for assessment of airway opening pressure without the need for low-flow insufflation. Crit Care. 2023 Jul 7;27(1):273. doi: 10.1186/s13054-023-04560-0. PMID 37420282
- [Background] Rodriguez Guerineau L, Vieira F, Rodrigues A, Reise K, Todd M, Guerguerian AM, Brochard L. Airway opening pressure maneuver to detect airway closure in mechanically ventilated pediatric patients. Front Pediatr. 2024 Feb 6;12:1310494. doi: 10.3389/fped.2024.1310494. eCollection 2024. PMID 38379913